CLINICAL TRIAL: NCT03465696
Title: A Priming Intervention to Increase Patient Willingness to Use Injectables for the Management of Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00049576
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
Keywords: psoriasis; biologics; treatment decision-making
MeSH Terms: conditions — Psoriasis | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group #1 (Control) (No Intervention): Group #1 (Control)
  Oral survey 1 will be administered and patients will be asked:
  Stelara® inhibits interleukin 23, one of the immune signaling molecules involved in psoriasis.
  How willing would you be to take Stelara® to treat your psoriasis, on a scale of (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing)
- Group #2 (Intervention) (Experimental): Group #2 (Intervention)
  Survey 2 will be administered, and patients will be asked the following primer:
  Stelara® inhibits interleukin 23, one of the immune signaling molecules involved in psoriasis. People who are born with a genetic deficiency in the immune signal interleukin-23 are generally healthy, but also have a LOWER risk of getting immune diseases like psoriasis.
  How willing would you be to take Stelara® to treat your psoriasis, on a scale of (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing)
  Interventions: Behavioral: Group #2 (Intervention)
- Group #3 (Intervention) (Experimental): Group #3 (Intervention)
  Survey 3 will be administered, and patients will be asked the following primer:
  Stelara® inhibits interleukin 23, one of the immune signaling molecules involved in psoriasis. People who are born with a genetic deficiency in the immune signal interleukin-23 are generally healthy, but also have a LOWER risk of getting immune diseases like psoriasis.
  What do you think would be the best way to describe this to a patient?
  1. Stelara® acts in an almost all-natural way to help control psoriasis.
  2. Stelara® blocks one of the genetic causes of psoriasis.
  3. Stelara® makes psoriasis better by blocking the overactive signal that gets the immune system out of balance
  4. Stelara® blocks interleukin-23, an important immune system signaling molecule involved in psoriasis
  How willing would you be to take Stelara® to treat your psoriasis, on a scale of (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing)
  Interventions: Behavioral: Group #3 (Intervention)

INTERVENTIONS:
Behavioral: Group #2 (Intervention) — Group #2 (Intervention)
  Survey 2 will be administered, and patients will be asked the following primer:
  Stelara® inhibits interleukin 23, one of the immune signaling molecules involved in psoriasis. People who are born with a genetic deficiency in the immune signal interleukin-23 are generally healthy, but also have a LOWER risk of getting immune diseases like psoriasis.
  How willing would you be to take Stelara® to treat your psoriasis, on a scale of (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing)
  Arms: Group #2 (Intervention)
Behavioral: Group #3 (Intervention) — Group #3 (Intervention)
  Survey 3 will be administered, and patients will be asked the following primer:
  Stelara® inhibits interleukin 23, one of the immune signaling molecules involved in psoriasis. People who are born with a genetic deficiency in the immune signal interleukin-23 are generally healthy, but also have a LOWER risk of getting immune diseases like psoriasis.
  What do you think would be the best way to describe this to a patient?
  1. Stelara® acts in an almost all-natural way to help control psoriasis.
  2. Stelara® blocks one of the genetic causes of psoriasis.
  3. Stelara® makes psoriasis better by blocking the overactive signal that gets the immune system out of balance
  4. Stelara® blocks interleukin-23, an important immune system signaling molecule involved in psoriasis
  How willing would you be to take Stelara® to treat your psoriasis, on a scale of (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing)
  Arms: Group #3 (Intervention)

SUMMARY:
Biologic medications have revolutionized the treatment of inflammatory diseases such as moderate-to-severe psoriasis. Though very effective with an excellent safety profile, patients may be apprehensive about choosing a biologic medication for a variety of reasons. The purpose of this research study is to learn more about patient's perception of certain psoriasis treatment options.

DETAILED DESCRIPTION:
The study will be conducted at the Wake Forest University Dermatology Clinic and on Amazon Mechanical Turk. Patients meeting the following characteristics will be eligible to participate: individuals diagnosed with psoriasis (ICD-9: 696.1) or a parent/caregiver of an individual diagnosed with psoriasis (ICD-9: 696.1). The study team will recruit 180 subjects for the study. Patients will be randomized to three survey groups.

Amazon Mechanical Turk, https://www.mturk.com/mturk/welcome, Amazon Mechanical Turk is an online crowdsourcing platform. The purpose of Mechanical Turk (MTurk) is to help people (participants) find paid tasks. In recent years MTurk had been extensively used in social science research.3 MTurk enables researchers to recruit participants to perform tasks such as filling out surveys, opinion polls, & cognitive psychological studies. Researchers advertise their studies on MTurk, and participants chose only those studies that interest them.

Amazon Turk had been extensively used by psychologists in the last few years for participant recruitment. Participants on Amazon Turk see a list of potential jobs (referred to as HITs) when they log into their MTurk account. The price is provided next to the name of the HIT along with the approximate length of time that the HIT will take. Participants are free to choose the HITs that they are interested in taking, from a long list of thousands of tasks. The name of our HIT will be "Treatment of Psoriasis - the patient's perspective". The survey takes approximately one minute to complete. Once participants click on the HIT, they will be taken directly to the survey (attached as supporting document) which provides further information about the study. The survey/study will be hosted on "Google forms, Survey monkey, Qualtrics or other survey form". MTurk rules state that participants can terminate the study by returning the HIT at any time, without any penalty.

Subjects will be randomized using SPSS version 24.0 or later into three groups and administered surveys querying willingness to use a biologic medication.

The surveyor will record patient responses in the study log if patient is recruited at the Wake Forest Dermatology Clinic. If recruited via MTurk, patient responses will be recorded through the MTurk log.

ELIGIBILITY:
Inclusion Criteria:

* Either diagnosed with psoriasis (ICD-9: 696.1) or a parent/caregiver of an individual diagnosed with psoriasis (ICD-9: 696.1).
* Subjects with a working knowledge of English.

Exclusion Criteria:

* Already on or previously failed management attempts with an IL-23 inhibitor including ustekinumab, guselkumab, risankizumab, or Tildrakizumab, amongst others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Oral Survey Responses | 12 months
  Oral survey responses, on a (1 = definitely willing, 2 = probably willing, 3 = probably not willing, 4 = definitely not willing) scale to take a treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No